CLINICAL TRIAL: NCT02383771
Title: Reversal of the Anti-platelet Effects of Ticagrelor in Healthy Persons and Patients With Coronary Artery Disease
Brief Title: Reversal of the Anti-platelet Effects of Ticagrelor
Acronym: REVERSAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chunjian Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2015-02-05; First posted 2015-03-09 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease
Keywords: Ticagrelor; Aspirin; Peri-operative treatment
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single Anti-platelet Treatment (Experimental): Ticagrelor
  Interventions: Drug: Ticagrelor
- Dual Anti-platelet Treatment (Experimental): Aspirin + Ticagrelor
  Interventions: Drug: Aspirin + Ticagrelor
- Control (Sham Comparator): No Drug
  Interventions: Drug: Control
- CAD undergoing PCI (Other): Patients with coronary artery disease undergoing percutaneous coronary intervention and receiving dual anti-platelet therapy (ticagrelor 90mg bid + aspirin 100mg daily)
  Interventions: Drug: Aspirin + Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — (Ticagrelor 90mg Bid) x 7days
  Other Names: Brilinta
  Arms: Single Anti-platelet Treatment
Drug: Aspirin + Ticagrelor — (Aspirin 100mg daily + Ticagrelor 90mg Bid) x 7days
  Other Names: Brilinta
  Arms: Dual Anti-platelet Treatment
Drug: Control — No Anti-platelet Therapy
  Arms: Control
Drug: Aspirin + Ticagrelor — Dual anti-platelet therapy (Aspirin 100mg daily + Ticagrelor 90mg Bid) after percutaneous coronary intervention (PCI)
  Other Names: Brilinta
  Arms: CAD undergoing PCI

SUMMARY:
The purpose of this study is to determine the proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of ticagrelor and aspirin in healthy persons and patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) and receiving ticagrelor.

DETAILED DESCRIPTION:
Reversal of the Anti-platelet Effects of Ticagrelor: REVERSAL study

The fatality of stent thrombosis (ST) in patients with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI) is approximately 50% and clopidogrel is an important anti-platelet drug for prevention of ST. CAD patients implanted with stent including bare metal stent (BMS) and drug eluting stent (DES) are recommended to receive dual anti-platelet treatment (DAPT), i.e. clopidogrel along with aspirin, for at least one year to reduce the incidence of ST by up-to-date guidelines. However, due to the variability of anti-platelet effect of clopidogrel, regular dose (75 mg daily) of clopidogrel administered cannot achieve enough inhibition of platelet aggregation in 20-30% of total patients, which is named as clopidogrel low responsiveness (CLR), and the morbidity of thrombosis (including) in CAD patients is still 10%.

Ticagrelor, a cyclopentyl-triazolo-pyrimidine, is a more potent adenosine diphosphate (ADP) receptor antagonist with faster onset and more significantly higher inhibition of platelet aggregation compared with clopidogrel and directly acts on P2Y12-ADP receptor in platelets without process of hepatic metabolism. In the PLATO study, ticagrelor plus reduced the remarkable incidence of cardiovascular events in patients with acute coronary syndrome (ACS) without significant higher incidence of major bleeding events compared with clopidogrel plus aspirin. Surprisingly, the incidence of death due to cardiovascular causes and the total fatality was decreased in patients with ticagrelor plus aspirin compared with those with clopidogrel plus aspirin. The results suggested the more benefit brought by ticagrelor, highlighting the wide use of it in the future.

Due to the potent anti-platelet effect of ticagrelor, more bleeding events may occur. Additionally, when facing the need for cardiac or non-cardiac operation, occurrence of life-threatening bleeding event or necessity of emergency operation, doctors may be confused of the treatment for the patients taking ticagrelor, of which the half-life period is 8-9 hours and it suggests the importance of studying the reversal of the anti-platelet effects of ticagrelor.

The primary objective of this study is to investigate the proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of aspirin and ticagrelor in healthy persons and patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) and receiving ticagrelor.

Study Population:

The investigators design two cohort studies, and plan to enroll 32 healthy volunteers in cohort 1 and 16 patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) and receiving dual anti-platelet therapy (ticagrelor 90mg bid + aspirin 100mg daily) for 7 days

Cohort 1:

Randomization:

A total of 32 healthy volunteers are planned to be enrolled and will be randomly divided into three groups: single anti-platelet treatment group (A group, 8 of 32), dual anti-platelet treatment group (B group, 8 of 32) and control group (C group, 16 of 32).

1. Single anti-platelet treatment group: (Ticagrelor 90mg bid) × 7 days
2. Dual anti-platelet treatment group: (Ticagrelor 90mg bid + Aspirin 100mg daily) × 7 days
3. Control group: No anti-platelet therapy

Inclusion criteria:

1. Healthy volunteers
2. Participants aged >18 years old

Exclusion criteria:

1. Allergy or intolerance to aspirin or ticagrelor;
2. Subjects at a high risk of bleeding (e.g. platelet count<100×10^9/L, history of peptic ulcer, hemoglobin<110g/L);
3. Subjects with bronchial asthma or chronic obstructive pulmonary disease;
4. Subjects with bradycardia (e.g. sick sinus syndrome, high-grade atrioventricular block, history of syncope with unproved uncorrelation with bradycardia);
5. Smokers;
6. Subjects with diabetes mellitus;
7. Subjects planning to be pregnancy;
8. Subjects with hepatic or renal dysfunction;
9. Subjects who have taken other anti-platelet drugs, non-steroidal anti-inflammatory drugs or proton pump inhibitors before scanning or need to take them during study period.

Blood collection and sample preparation

Venous blood samples are collected by venipuncture into two 4.5-mL draw BD vacutainer tubes containing 0.105M buffered sodium citrate (3.2%) at 08.00 hours in the morning before taking the agent and after the last dose of the study drug. Platelet-rich plasma (PRP) from subjects in A group is mixed with increasing proportions of that in C group, with one untreated subject serving as the control for one treated subject. The proportion of control platelets mixed with inhibited platelets is calculated based on platelet numbers, starting at 10% and increasing by 10% increments. So as the PRP in B group.

Test:

1. Before taking the agent:

   1. ADP-induced platelet aggregation: light transmittance aggregation (LTA) in response to 5μM ADP
   2. Arachidonic acid (AA)-induced platelet aggregation: LTA in response to 1mM AA
2. After 7-day medication:

   1. ADP-induced platelet aggregation: LTA in response to 5μM ADP
   2. AA-induced platelet aggregation: LTA in response to 1mM AA
   3. ADP-induced platelet aggregation of mixed sample: LTA in response to 5μM ADP
   4. AA-induced platelet aggregation of mixed sample: LTA in response to 1mM AA

Primary end points:

1. Reversal of the platelet inhibitory effects of antiplatelet therapy Proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of antiplatelet therapy in healthy volunteers

Secondary end points:

1. Inhibition of platelet aggregation (IPA) in response to 5μM ADP determined by light transmittance aggregometer (LTA) after 7-day ticagrelor administration

Safety issue: No

Cohort 2:

A total of 16 patients with diagnosed coronary artery disease who have undergone percutaneous coronary intervention (PCI) and have received dual anti-platelet therapy (ticagrelor 90mg bid + aspirin 100mg daily) for 7 days is planned to be enrolled.

Inclusion Criteria:

1. Subjects with diagnosed coronary artery disease undergoing percutaneous coronary intervention (PCI);
2. Subjects who have received dual anti-platelet therapy (ticagrelor 90mg bid + aspirin 100mg daily) for 7 days;

Exclusion Criteria:

1. Subjects at a high risk of bleeding (e.g. platelet count<100×10^9/L, history of peptic ulcer, hemoglobin<110g/L);
2. Subjects with anemia;
3. Smokers
4. Subjects planning to be pregnancy;
5. Subjects with hepatic or renal dysfunction;
6. Subjects who have taken other anti-platelet drugs, non-steroidal anti-inflammatory drugs or proton pump inhibitors before scanning or need to take them during study period.

Sample test for fresh platelet saved in blood bank

Function of platelet aggregation, platelet count, pH value and metabolic products (including PO2, PCO2, blood glucose, lactate, bicarbonate, sodium, potassium and chloride) are measured in fresh platelet sample preserved in blood bank for 1, 2, 3, 4, and 5 days respectively.

Blood collection and sample preparation for patients

Venous blood samples are collected by venipuncture into two 4.5-mL draw BD vacutainer tubes containing 0.105M buffered sodium citrate (3.2%) at 08.00 hours in the morning after taking the medicine. Platelet-rich plasma (PRP) from participants is mixed with increasing proportions of that extracted from fresh platelet sample reserved in blood bank for one day as the control for each treated subject. The proportion of control platelets mixed with inhibited platelets is calculated based on platelet numbers, starting at 10% and increasing by 10% increments. So as the PRP mixed with fresh platelet sample preserved for four days.

Test for sample from patients

1. Before mixture:

   1. ADP-induced platelet aggregation: light transmittance aggregation (LTA) in response to 5μM ADP
   2. Arachidonic acid (AA)-induced platelet aggregation: LTA in response to 1mM AA
2. After mixture:

   1. ADP-induced platelet aggregation: LTA in response to 5μM ADP
   2. AA-induced platelet aggregation: LTA in response to 1mM AA

Primary end points:

1. Reversal of the platelet inhibitory effects of antiplatelet therapy Proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of antiplatelet therapy in patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) and receiving ticagrelor

Secondary end points:

1. Relationship between function of platelet aggregation and the time of saving fresh platelet.

Safety issue: No

ELIGIBILITY:
Cohort 1:

Inclusion Criteria:

* Healthy volunteers;
* Subjects aged >18 years old;

Exclusion Criteria:

* Allergy or intolerance to aspirin or ticagrelor;
* Subjects at a high risk of bleeding (e.g. platelet count<100×10^9/L, history of peptic ulcer, hemoglobin<110g/L);
* Subjects with anemia;
* Subjects with bronchial asthma or chronic obstructive pulmonary disease;
* Subjects with bradycardia (e.g. sick sinus syndrome, high-grade atrioventricular block, history of syncope with unproved uncorrelation with bradycardia);
* Smokers;
* Subjects with diabetes mellitus;
* Subjects planning to be pregnancy;
* Subjects with hepatic or renal dysfunction;
* Subjects who have taken other anti-platelet drugs, non-steroidal anti-inflammatory drugs or proton pump inhibitors before scanning or need to take them during study period.

Cohort 2:

Inclusion Criteria:

* Subjects with diagnosed coronary artery disease undergoing percutaneous coronary intervention (PCI);
* Subjects who have received dual anti-platelet therapy (ticagrelor 90mg bid + aspirin 100mg daily) for 7 days;

Exclusion Criteria:

* Subjects at a high risk of bleeding (e.g. platelet count<100×10^9/L, history of peptic ulcer, hemoglobin<110g/L);
* Subjects with anemia;
* Smokers
* Subjects planning to be pregnancy;
* Subjects with hepatic or renal dysfunction;
* Subjects who have taken other anti-platelet drugs, non-steroidal anti-inflammatory drugs or proton pump inhibitors before scanning or need to take them during study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Reversal of the platelet inhibitory effects of antiplatelet therapy in healthy volunteers | 7 days after randomization
  Proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of antiplatelet therapy
Reversal of the platelet inhibitory effects of antiplatelet therapy in patients | 7 days after percutaneous coronary intervention
  Reversal of the platelet inhibitory effects of antiplatelet therapy Proportion of untreated donor platelets required to fully reverse the platelet inhibitory effects of antiplatelet therapy in patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) and receiving ticagrelor

SECONDARY OUTCOMES:
Inhibition of platelet aggregation in response to AA or ADP | 7 days after randomization
  Inhibition of platelet aggregation (IPA) in response to 5μM ADP determined by light transmittance aggregometer (LTA) after 7-day ticagrelor administration
Change of ADP-induced platelet aggregation in platelets saved in blood bank due to the saving time | 5 days after fresh platelet collected and stored in blood bank
  How the ADP-induced platelet aggregation in platelets saved in blood bank changes due to the saving time

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] Kushner FG, Hand M, Smith SC Jr, King SB 3rd, Anderson JL, Antman EM, Bailey SR, Bates ER, Blankenship JC, Casey DE Jr, Green LA, Hochman JS, Jacobs AK, Krumholz HM, Morrison DA, Ornato JP, Pearle DL, Peterson ED, Sloan MA, Whitlow PL, Williams DO. 2009 focused updates: ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction (updating the 2004 guideline and 2007 focused update) and ACC/AHA/SCAI guidelines on percutaneous coronary intervention (updating the 2005 guideline and 2007 focused update) a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2009 Dec 1;54(23):2205-41. doi: 10.1016/j.jacc.2009.10.015. No abstract available. PMID 19942100
- [Background] Nguyen TA, Diodati JG, Pharand C. Resistance to clopidogrel: a review of the evidence. J Am Coll Cardiol. 2005 Apr 19;45(8):1157-64. doi: 10.1016/j.jacc.2005.01.034. PMID 15837243
- [Background] Trenk D, Hochholzer W, Fromm MF, Chialda LE, Pahl A, Valina CM, Stratz C, Schmiebusch P, Bestehorn HP, Buttner HJ, Neumann FJ. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drug-eluting or bare-metal stents. J Am Coll Cardiol. 2008 May 20;51(20):1925-34. doi: 10.1016/j.jacc.2007.12.056. PMID 18482659
- [Background] Ellis KJ, Stouffer GA, McLeod HL, Lee CR. Clopidogrel pharmacogenomics and risk of inadequate platelet inhibition: US FDA recommendations. Pharmacogenomics. 2009 Nov;10(11):1799-817. doi: 10.2217/pgs.09.143. PMID 19891556
- [Background] Chong AY, So DY. Ticagrelor for the treatment of peripheral arterial disease. Expert Opin Investig Drugs. 2014 Dec;23(12):1737-43. doi: 10.1517/13543784.2014.974803. Epub 2014 Nov 6. PMID 25376000
- [Background] Solbeck S, Meyer MA, Johansson PI, Meyer AS, Cotton BA, Stensballe J, Schott U, Ostrowski SR. Monitoring of dabigatran anticoagulation and its reversal in vitro by thrombelastography. Int J Cardiol. 2014 Oct 20;176(3):794-9. doi: 10.1016/j.ijcard.2014.07.084. Epub 2014 Aug 4. PMID 25156858
- [Background] Montalescot G, van 't Hof AW, Lapostolle F, Silvain J, Lassen JF, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Goodman SG, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Zeymer U, Stibbe O, Ecollan P, Heutz WM, Swahn E, Collet JP, Willems FF, Baradat C, Licour M, Tsatsaris A, Vicaut E, Hamm CW; ATLANTIC Investigators. Prehospital ticagrelor in ST-segment elevation myocardial infarction. N Engl J Med. 2014 Sep 11;371(11):1016-27. doi: 10.1056/NEJMoa1407024. Epub 2014 Sep 1. PMID 25175921
- [Background] Gurbel PA, Antonino MJ, Tantry US. Recent developments in clopidogrel pharmacology and their relation to clinical outcomes. Expert Opin Drug Metab Toxicol. 2009 Aug;5(8):989-1004. doi: 10.1517/17425250903107772. PMID 19575629
- [Background] Cannon CP, Harrington RA, James S, Ardissino D, Becker RC, Emanuelsson H, Husted S, Katus H, Keltai M, Khurmi NS, Kontny F, Lewis BS, Steg PG, Storey RF, Wojdyla D, Wallentin L; PLATelet inhibition and patient Outcomes Investigators. Comparison of ticagrelor with clopidogrel in patients with a planned invasive strategy for acute coronary syndromes (PLATO): a randomised double-blind study. Lancet. 2010 Jan 23;375(9711):283-93. doi: 10.1016/S0140-6736(09)62191-7. Epub 2010 Jan 13. PMID 20079528
- [Background] Li C, Hirsh J, Sloane D, Liang Y, Bai J, Paikin J, Johnston MA, DeBeer J, Eikelboom JW. Aspirin response variability after major orthopedic surgery. Thromb Res. 2012 Aug;130(2):216-20. doi: 10.1016/j.thromres.2012.04.006. Epub 2012 May 9. PMID 22575418
- [Background] Teng R, Butler K. Pharmacokinetics, pharmacodynamics, tolerability and safety of single ascending doses of ticagrelor, a reversibly binding oral P2Y(12) receptor antagonist, in healthy subjects. Eur J Clin Pharmacol. 2010 May;66(5):487-96. doi: 10.1007/s00228-009-0778-5. Epub 2010 Jan 21. PMID 20091161
- [Background] Li C, Hirsh J, Xie C, Johnston MA, Eikelboom JW. Reversal of the anti-platelet effects of aspirin and clopidogrel. J Thromb Haemost. 2012 Apr;10(4):521-8. doi: 10.1111/j.1538-7836.2012.04641.x. PMID 22268852
- [Background] Hobl EL, Derhaschnig U, Firbas C, Schoergenhofer C, Schwameis M, Jilma B. Reversal strategy in antagonizing the P2Y12 -inhibitor ticagrelor. Eur J Clin Invest. 2013 Dec;43(12):1258-61. doi: 10.1111/eci.12168. Epub 2013 Sep 23. PMID 24112116
- [Background] Storey RF, Bliden KP, Ecob R, Karunakaran A, Butler K, Wei C, Tantry U, Gurbel PA. Earlier recovery of platelet function after discontinuation of treatment with ticagrelor compared with clopidogrel in patients with high antiplatelet responses. J Thromb Haemost. 2011 Sep;9(9):1730-7. doi: 10.1111/j.1538-7836.2011.04419.x. PMID 21707911
- [Background] Coelho MJ, Monteiro Tde C, Vasquez FG, Silva KL, Dos Santos KS, de Oliveira VM, Cavalcante Fde O. Platelet aggregation and quality control of platelet concentrates produced in the Amazon Blood Bank. Rev Bras Hematol Hemoter. 2011;33(2):110-4. doi: 10.5581/1516-8484.20110030. PMID 23284257
- [Background] Shams Hakimi C, Hesse C, Wallen H, Boulund F, Grahn A, Jeppsson A. In vitro assessment of platelet concentrates with multiple electrode aggregometry. Platelets. 2015;26(2):132-7. doi: 10.3109/09537104.2014.898141. Epub 2014 Jul 7. PMID 24999542